CLINICAL TRIAL: NCT03623711
Title: A Prediction Study of Multiple Indexes of the Effect of Different Mechanisms of Antidepressants Treatment on Depression
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuqi Cheng (Other)
Responsible Party: Sponsor-Investigator, Yuqi Cheng, Associate professor, Kunming Medical University
Organization: Kunming Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81660237
Record Dates: First submitted 2017-07-14; First posted 2018-08-09 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Major Depressive Disorder; Depression, Unipolar
Keywords: major depressive disorder; Magnetic Resonance Imaging; Antidepressant Treatment
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder | interventions — Escitalopram; Duloxetine Hydrochloride; Bupropion

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Escitalopram group (Experimental): including 50 patients, dosage:start 10mg/day and last 2 weeks,we assess the HAMD score at the end of 2 weeks, if the reduction rate of HAMD less than 20% relative to baseline, the dosage add to 20mg/day and last to the end of 12 week. but if the reduction rate of HAMD more than 20% relative to baseline, the investigators will continue to use current dosage until the end of 12 week.
  Interventions: Drug: Escitalopram
- Duloxetine group (Experimental): including 50 patients, dosage:start 30mg/day and last 2 weeks,we assess the HAMD score at the end of 2 weeks, if the reduction rate of HAMD less than 20% relative to baseline, the dosage add to 60mg/day and last to the end of 12 week. but if the reduction rate of HAMD more than 20% relative to baseline,the investigators will continue to use current dosage until the end of 12 week.
  Interventions: Drug: Duloxetine
- Bupropion group (Experimental): including 50 patients, dosage:start 75mg/day and last 2 weeks,we assess the HAMD score at the end of 2 weeks, if the reduction rate of HAMD more than 20% relative to baseline, the investigators will continue to use current dosage until the end of 12 week.if the reduction rate of HAMD less than 20% relative to baseline, the dosage add to 150mg/day and last 2 weeks, the investigators assess the HAMD score again, if the reduction rate of HAMD more than 20% relative to baseline, the investigators will continue to use current dosage until the end of 12 week, but if the reduction rate of HAMD still less than 20% relative to baseline, the participants would withdraw.
  Interventions: Drug: Bupropion
- Healthy control (Placebo Comparator): 50 age-, gender-,education level- and handedness matched healthy control would recruit by an advertisement in the local community and school, and excluding ① with a severe physical disease and/or neurological disease, ②with substance abuse, ③ with a history of brain injury, ④ inability to undergo a MRI scan.
  Interventions: Other: Healthy control

INTERVENTIONS:
Drug: Escitalopram — participants take escitalopram tablets based on their severity of depression (10-20mg/day) at least for 12 weeks.
  Other Names: Lexapro
  Arms: Escitalopram group
Drug: Duloxetine — participants take Duloxetine capsule based on their severity of depression (60mg/day) at least for 12 weeks.
  Other Names: cymbalta
  Arms: Duloxetine group
Drug: Bupropion — participants take Bupropion tablets based on their severity of depression (75-300mg/day) at least for 12 weeks.
  Other Names: bupropion hydrochloride tablets
  Arms: Bupropion group
Other: Healthy control — Healthy control take placebo tablets
  Other Names: placebo tablets
  Arms: Healthy control

SUMMARY:
Antidepressants is the primary treatment for depression, but only less than 50% of the patients get clinical remission. There is no objective markers to select antidepressants for clinical treatment . Clinical choose usually use experience and waste a lot of time, even the patients cannot be treated timely and effectively. The investigators found that the later antidepressant effect for 8 weeks is related with early brain functional response. Present prospectively drug treatment and follow-up study intends to adopt pharmacological imaging research methods to detect the brain function or structure change of three different mechanisms of antidepressant drugs, selective serotonin reuptake inhibitors (SSRIs, escitalopram), serotonin and norepinephrine reuptake inhibitors (SNRIs, duloxetine), norepinephrine and dopamine reuptake inhibitors (NDRIs, bupropion) in depression patients. Brain functional or structural magnetic resonance imaging data were collected at baseline, 1 days, 14 days and 12 weeks after treatment. The investigators want to observe the changes of brain functional networks and structure at different time points, acute and chronic treatment induced during drug treatment. Combined with the blood concentration detection, symptom change, cognitive function tests, the investigators also hope to determine the different mechanisms of drug efficacy of antidepressants with different mechanisms. The second aim is to explore different mechanisms of brain function for effective or ineffective drug response. The results of the study will help to further explain the mechanism of different antidepressants, to facilitate the development of early indicators for drug efficacy and individual treatment decision.

DETAILED DESCRIPTION:
about 150 depression patients were divided into three subgroups, for each group was treated by one antidepressant eg.escitalopram,duloxetine,bupropion.Brain magnetic resonance imaging data were conducted for all patients at baseline, 1 days, 14 days and 12 weeks after treatment. The blood concentration detection, symptom change, cognitive function tests were also conducted. combined with these results the investigators aim to determine the different mechanisms of drug efficacy of antidepressants with different mechanisms and to explore different mechanisms of brain function for effective or ineffective drug response

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual (DSM)-IV Major Depression or Dysthymia
* Age 18-60
* Physically healthy
* The score of Hamilton Depression Rating Scale (HAMD)≥18 points
* Drug-free

Exclusion Criteria:

* Body metal (e.g., wire stitches, screws in bones, stainless steel hips)
* History of Psychosis or Epilepsy
* Current (past six months) Substance Use Disorder (illicit drugs and/or alcohol)
* Bipolar I
* Need for wash-out from effective treatment in order to participate
* Pregnant or breastfeeding
* High suicide risk
* Currently taking (within 2 weeks; 4 weeks for Fluoxetine) antidepressants
* have received regular treatment of electric convulsions, repetitive transcranial magnetic stimulation (rTMS), or systematic psychotherapy within three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
change of functional magnetic resonance imaging (fMRI) after medication | at baseline, 1 days, 14 days and 12 weeks after treatment
  change of fMRI after medication

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided